CLINICAL TRIAL: NCT04851613
Title: A Phase Ib/III Study to Evaluate the Efficacy and Safety of Afuresertib Plus Fulvestrant in Patients With Locally Advanced or Metastatic HR+/HER2- Breast Cancer Who Failed Standard of Care Therapies
Brief Title: Study to Evaluate Efficacy & Safety of Afuresertib Plus Fulvestrant in Patients With Locally Advanced or Metastatic HR+/HER2- Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laekna Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAE205INT3101
Record Dates: First submitted 2021-04-13; First posted 2021-04-20 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — afuresertib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Phase I: Single-arm, open-label study to evaluate efficacy, safety, tolerability, PK of the therapy with afuresertib plus fulvestrant. Phase III: A multi-center, randomized, double-blind, placebo-controlled study to assess efficacy and safety of afuresertib/placebo plus fulvestrant in patients with HR+/HER2- locally advanced or metastatic BC who have failed 1 to 2 prior lines of ET with/without a CDK4/6 inhibitor (up to 1 therapy), or chemotherapy (up to 1 chemotherapy).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase I: Afuresertib and Fulvestrant Safety Run In (Experimental): Phase I: Safety run-in Cycle 1 (a cycle is 28 days) will be performed in the first 6 patients of the phase Ib. Combination regimens during the safety run-in period are: afuresertib 125 mg QD (once daily) + fulvestrant 500 mg Intra Muscular (IM) on Day 1, 15 of Cycle 1, and on Day 1 of the subsequent 28-day cycles.
  Interventions: Drug: Afuresertib
- Phase I: Afuresertib and Fulvestrant (Experimental): Phase I: Combination regimens are: afuresertib 125 mg QD (once daily) + fulvestrant 500 mg Intra Muscular (IM) on Day 1, 15 of Cycle 1, and on Day 1 of the subsequent 28-day cycles.
  Interventions: Drug: Afuresertib
- Phase III: afuresertib combined with fulvestrant (experimental arm) (Experimental): Phase III: afuresertib 125mg QD combined with fulvestrant 500mg Q4W (D1, 15 in cycle 1)
  Interventions: Drug: Afuresertib
- Phase III: placebo combined with fulvestrant (control arm) (Placebo Comparator): PhaseIII：placebo combined with fulvestrant 500mg Q4W (D1, 15 in cycle 1)
  Interventions: Drug: Afuresertib/placebo

INTERVENTIONS:
Drug: Afuresertib — The starting doses of the combination therapy are afuresertib 125 mg PO, QD plus fulvestrant 500 mg IM, D1, 15 in the first cycle and afuresertib 125 mg PO, QD plus fulvestrant 500 mg IM, D1 Q4W in the subsequent cycles
  Other Names: Fulvestrant
  Arms: Phase I: Afuresertib and Fulvestrant; Phase I: Afuresertib and Fulvestrant Safety Run In; Phase III: afuresertib combined with fulvestrant (experimental arm)
Drug: Afuresertib/placebo — afuresertib/placebo 125mg QD combined with fulvestrant 500mg Q4W (D1, 15 in cycle 1)
  Other Names: Fulvestrant
  Arms: Phase III: placebo combined with fulvestrant (control arm)

SUMMARY:
Study LAE205INT3101 is a Phase Ib/III study to evaluate the efficacy and safety of the combination therapy with afuresertib plus fulvestrant (afuresertib/placebo plus fulvestrant in Phase III) in patients with HR+/HER2- breast cancer who have failed 1 to 2 prior lines of endocrine therapy, and/or CDK4/6 inhibitor (up to 1 therapy), and/or chemotherapy (up to 1 chemotherapy) as described in the inclusion criteria.

DETAILED DESCRIPTION:
Eligible patients for this study must have either (1) progressive disease whilst receiving an endocrine therapy (AI or a SERM), and/or a CDK4/6 inhibitor for locally advanced or metastatic disease; or (2) relapsed with metastatic disease whilst receiving an ET (AI or SERM), and/or a CDK4/6 inhibitor, and/or chemotherapy in adjuvant setting. No more than 2 prior lines of systemic treatments for locally advanced or metastatic disease are allowed for this study, including 1-2 prior lines of endocrine therapy, with/without CDK4/6 inhibitor (up to 1 therapy), and/or chemotherapy (up to 1 therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients must be ≥ 18 years of age on the day of signing the informed consent and be able to provide written informed consent for the study.
2. Patients with histologically or cytologically confirmed HR+/HER2- Breast Cancer characterized by the absence of HER2 expression and the presence of ER with/without PR expression.
3. Female patients may be post-menopausal, pre-menopausal or peri-menopausal. Male and Pre- and peri-menopausal females may be enrolled if continuously treated with ovarian suppression therapy (use LHRHa at least starting from C1D1) for the duration of study participation.
4. Before enrollment, patients who have undergone anti-cancer treatment must have a washout period of 4 weeks or 5 half-lives, whichever comes earlier.
5. HR+/HER2- BC patients must meet all the following criteria to join this study:

   1. Relapsed locally advanced (LABC) or metastatic (mBC) disease; AND
   2. Have received 1 to 2 prior lines of systemic treatments for LABC or mBC(at least one line was ET). If disease relapse during adjuvant therapy or relapse within 12 months from completion of adjuvant endocrine therapy, the adjuvant therapy will be counted as 1 line), including:

   i. Endocrine therapies including AIs and/or SERMs (1 or 2 lines) with or without a CDK4/6 inhibitor (up to 1 therapy); OR ii. A chemotherapy (monotherapy or combination therapy, at most 1 line only), with 1 additional line of endocrine therapy .
6. For phase Ib part, patients must have at least one lesion that meets the definition of measurable disease by RECIST 1.1 criteria; for phase III, have measurable disease and/or at least 1 lytic or mixed (lytic + sclerotic) bone lesion that can be assessed by RECIST 1.1 criteria; patients with sclerotic/osteoblastic bone lesions only in the absence of measurable disease are not eligible (Appendix 2).
7. In the Phase Ib part, Patients must provide informed consent for the procedures and the tests for PIK3CA/AKT/PTEN alterations and ESR1 mutations. The biomarkers will be tested retrospectively by gene sequencing tests using archival tumor sample (preferably within 18 months/78 weeks) or from peripheral blood or from a tumor biopsy sample. Formalin-fixed, paraffin embedded (FFPE) tissue blocksare preferred. In phase III, blood sample is mandatory for this test.
8. In Phase III, subjects need to provide blood sample during the screening period for PIK3CA/AKT1/PTEN test, which will be conducted in the central laboratory. Only patients with PIK3CA/AKT1/PTEN alterations could include.
9. Patients with an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
10. Patients who have adequate organ function as defined.
11. Patients without a pre-existing diagnosis of diabetes mellitus (DM) who have a fasting glucose ≤ 126 mg/dL (or ≤ 7.0 mmol/L); or patients with type 2 diabetes who have a fasting glucose ≤ 167 mg/dL (or ≤ 9.3 mmol/L) AND glycosylated hemoglobin (HbA1c) ≤ 8%. Patients with DM type 1 or patients with DM type 2 requiring insulin or ≥21 anti-abetic medications for glycemic control are excluded.
12. Patients with a life expectancy of 24 weeks or more based on investigator's assessment.
13. Patients who have recovered from adverse events associated with pre-study medical, radiation and surgical treatments to ≤ Grade 1, excluding stable symptoms (e.g., alopecia, peripheral sensory neuropathy, skin hyperpigmentation, dysgeusia, etc.).
14. Female patients of childbearing potential must have a negative pretreatment serum pregnancy test.
15. Female patients of childbearing potential must agree to use effective contraception from enrollment to 1 year after discontinuation from the last dose of this study treatment.
16. Patients who are able to swallow and retain oral medication and without gastrointestinal diseases to interfere with drug absorption.
17. Patients must have no contraindications to fulvestrant.

Exclusion Criteria:

1. Patients who had a recent major surgery that required hospitalization for longer than 48 hours (< 8 weeks from scheduled treatment starting date) or have used IV antibiotics for the treatment of systemic infection (< 2 weeks from scheduled treatment starting date).
2. Patients who have additional known malignancies that are progressing or have required active treatments within 3 years of scheduled treatment starting date. (Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, that have undergone potentially curative therapy are not excluded).
3. Patients who have a history of seizure or conditions that may predispose them to seizure and require anti-epileptic medications, or patients who have brain arteriovenous malformation, or intracranial masses that are causing edema or clinical symptoms.
4. Patients who have known active CNS metastases and/or carcinomatous meningitis. (Note: Patients with previously treated brain metastases may participate provided that they are radiologically stable (i.e., without evidence of progression for at least 4 weeks by repeated imaging performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to schedule treatment starting date.
5. Patients who had prior treatment with fulvestrant or other selective estrogen receptor degraders (SERDs), or any PI3K/AKT/mTOR inhibitors, or any CDK4/6 inhibitors in phase I, II study.
6. Patients who had the following conditions within 6 months (26 weeks) of scheduled treatment starting date: New York Heart Association congestive heart failure classification III to IV, unstable angina, myocardial infarction, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or serious cardiac arrhythmia associated with significant cardiovascular impairment as determined by the investigator.
7. Patients with QT interval corrected by the Frederica's correction formula (QTcF) > 470 msec(average value), unless the prolonged QT interval is due to (right or left) bundle branch block and/or pacemaker rhythm. If wide QRS complex is present, cardiology consultation is required to assess the risk for Torsade de Pointes. Note: QTcF = QT/(RR^0.33) .
8. Patients who have uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg under anti-hypertensive treatment). Note: Patients with a history of hypertension are allowed, provided that blood pressure is controlled to within these limits by anti-hypertensive treatment.
9. Patients with active Hepatitis B infection [defined as HBsAg (+) and HBV-DNA ≥ 200 IU/ml (1000 copy/ml)] or active Hepatitis C virus [defined as HCV antibody positive and HCV RNA (qualitative) test positive].
10. Patients with known HIV seropositivity who has 1 of the following:

    1. Not receiving highly active antiretroviral therapy
    2. Receiving antiretroviral therapy that may interfere with the study drug (consult the Sponsor/Medical Monitor for review of medication prior to enrollment)
    3. CD4 count < 350 based on a test within 3 months of the screening visit
    4. An acquired immunodeficiency syndrome-defining opportunistic infection within 6 months (26 weeks) of the start of study screening
11. Patients who have a history or current evidence of any condition, therapy, or laboratory abnormality that in the opinion of the investigator, might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate.
12. Patients who have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
13. Patients who are receiving medications that are sensitive substrates of CYP3A4, OATP1B1, or BCRP with low therapeutic index. Please see related section for a list of these prohibited medications.
14. Patients who are currently pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 1 year after the last dose of study treatment.
15. Patients who have known cirrhosis with a Child-Pugh status of B and C.
16. Patients who are ineligible for endocrine therapy (e.g., visceral crisis, inflammatory breast cancer, uncontrolled pleural or abdominal fluid drainage ≥4 times within one month before planned administration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Overall Response Rate (ORR) based on RECIST 1.1 | Phase I: Change from Baseline beginning at Cycle 3 Day 1 and then every 8 weeks × 40 weeks then every 3 months through study completion, an average of 1 year (each cycle is 28 days)
  Phase I: Anti-tumor activity of the combination therapy with afuresertib plus fulvestrant in patients with HR+/HER2- BC
Phase III: Progression Free Survival (PFS) based on RECIST 1.1, as assessed by investigators | Phase III:Change from Baseline beginning at Cycle 3 Day 1 and then every 8 weeks for the first 12 months, then every 3 months through study completion
  Phase III:To assess the anti-tumor activity of the combination therapy with afuresertib plus fulvestrant versus placebo plus fulvestrant in patients with PIK3CA/AKT1/PTEN alterations HR+/HER2- BC who have failed 1 to 2 prior lines of ET with/without a Phase III: CDK4/6 inhibitor (up to 1 therapy), or chemotherapy (up to 1 chemotherapy)

SECONDARY OUTCOMES:
Phase I: Duration of Response (DOR) based on RECIST 1.1 | Phase I: Change from Baseline beginning at Cycle 3 Day 1 and then every 8 weeks x 40 weeks then every 3 months through study completion, an average of 1 year (each cycle is 28 days)
  Phase I: Anti-tumor activity of the combination therapy with afuresertib plus fulvestrant in patients with HR+/HER2- BC
Phase I: Clinical rate of benefit (CBR) based on RECIST 1.1 | Phase I: Change from Baseline beginning at Cycle 3 Day 1 and then every 8 weeks x 40 weeks then every 3 months through study completion, an average of 1 year (each cycle is 28 days)
  Phase I: Anti-tumor activity of the combination therapy with afuresertib plus fulvestrant in patients with HR+/HER2- BC
Phase I: Best Overall Response (BOR) based on RECIST 1.1 | Phase I: Change from Baseline beginning at Cycle 3 Day 1 and then every 8 weeks x 40 weeks then every 3 months through study completion, an average of 1 year (each cycle is 28 days)
  Phase I: Anti-tumor activity of the combination therapy with afuresertib plus fulvestrant in patients with HR+/HER2- BC
Phase I: Progression Free Survival (PFS) based on RECIST 1.1 | Phase I: After Cycle 3 Day 1 and then every 8 weeks x 40 weeks then every 3 months through study completion, an average of 1 year (each cycle is 28 days)
  Phase I: Anti-tumor activity of the combination therapy with afuresertib plus fulvestrant in patients with HR+/HER2- BC
Phase I: Pharmacokinetics- Time to Maximum Concentration (T-Max) | Phase I: Assessed on Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
  Phase I: Time to peak level of afuresertib
Phase I: Pharmacokinetics- Area Under the Curve (AUC) | Assessed on Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
  Area under the curve of afuresertib
Phase I: Frequency and severity of Adverse Events (AEs) | Phase I: Through study completion for an average of 12 months
  Phase I: findings on physical examination, ECG, vital signs, and reports of the laboratory results based on the CTCAE v5.0
Phase III: Progression Free Survival (PFS) based on RECIST 1.1, as assessed by BICR | Phase III:Change from Baseline beginning at Cycle 3 Day 1 and then every 8 weeks for the first 12 months then every 3 months through study completion
  Phase III: Anti-tumor activity of the combination therapy with afuresertib plus fulvestrant in patients with HR+/HER2- BC
Phase III：Frequency and severity of Adverse Events (AEs) | Phase III：Through study completion
  Phase III：findings on physical examination, ECG, vital signs, and reports of the laboratory results based on the CTCAE v5.0
Phase III：Pharmacokinetics- Time to Maximum Concentration (T-Max) | Assessed on Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
  Time to peak level of afuresertib
Phase III：Pharmacokinetics- Area Under the Curve (AUC) | Assessed on Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
  Area under the curve of afuresertib

CONTACTS AND LOCATIONS:
Overall Officials: Wenyue Ma, Study Director — Laekna Limited
Locations (55):
- United States (6):
  - Providence St. Johns Health Center, Santa Monica, California
  - Piedmont Cancer Institute, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Vermont, Burlington, Vermont
  - Virginia Cancer Specialists, Fairfax, Virginia
- China (49):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital (PUMCH), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen Memorial Hospital，Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang cancer hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir-run shaw Hospital Zhejiang University of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Ningbo Li Huili Hospital, Ningbo, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang

REFERENCES:
- [Derived] Zhang P, Sun T, Wang Y, Li W, Tong Z, Phadke S, Feinstein T, Ma W, Guo P, Zhang M, Yue Y, Xu B. Afuresertib plus fulvestrant for pretreated HR-positive, HER2-negative, advanced breast cancer: a phase Ib trial. Nat Commun. 2026 Feb 6. doi: 10.1038/s41467-026-69225-2. Online ahead of print. PMID 41651834